CLINICAL TRIAL: NCT03203876
Title: A Phase 1 Study of the Safety and Pharmacokinetics of Anti-KIR Monoclonal Antibody (Lirilumab, BMS-986015) in Combination With Anti-PD-1 Monoclonal Antibody (Nivolumab,BMS-936558) or in Combination With Nivolumab and Anti-CTLA-4 Monoclonal Antibody (Ipilimumab, BMS-734016) in Advanced and/or Metastatic Solid Tumors
Brief Title: A Safety Study of Lirilumab in Combination With Nivolumab or in Combination With Nivolumab and Ipilimumab in Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA223-030
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — lirilumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part One Combination Therapy (Experimental): Lirilumab and Nivolumab
  Interventions: Biological: Lirilumab; Biological: Nivolumab
- Part 2 Combination Therapy (Experimental): Lirilumab, Nivolumab and Ipilimumab
  Interventions: Biological: Lirilumab; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Lirilumab — Specified dose on specified days
  Other Names: BMS-986015
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy
  Arms: Part 2 Combination Therapy

SUMMARY:
The purpose of this study is to determine whether lirilumab in combination with nivolumab or in combination with nivolumab and ipilimumab is safe in the treatment of advanced and/or metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

* Participants must have histologic or cytologic confirmation of a solid malignancy that is advanced (metastatic and/or unresectable)
* Presence of at least 1 lesion with measurable disease as defined by response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) criteria for response assessment
* The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Participants with untreated central nervous system (CNS) metastases
* Participants with an active, known, or suspected autoimmune disease
* Uncontrolled or significant cardiovascular disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab
Incidence of adverse events (AEs) | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab
Incidence of serious adverse events (SAEs) | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab
Incidence of death | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab
Frequency of laboratory test toxicity grade shifting from baseline | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab
Incidence of AEs leading to discontinuation | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab

SECONDARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab and ipilimumab
Incidence of adverse events (AEs) | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab and ipilimumab
Incidence of serious adverse events (SAEs) | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab and ipilimumab
Incidence of death | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab and ipilimumab
Frequency of laboratory test toxicity grade shifting from baseline | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab and ipilimumab
Maximum serum observed concentration (Cmax) | Up to two years
  To characterize the Pharmacokinetic (PK) of lirilumab given in combination with nivolumab
Time of maximum observed serum concentration (Tmax) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration [AUC(0-T)] | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Trough observed serum concentration (Ctrough) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Area under the serum concentration-time curve in one dosing interval [AUC(TAU)] | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Clearance (CL) | Up to two years
  To characterize the PK and immunogenicity of lirilumab given in combination with nivolumab
Volume of distribution at steady state (Vss) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Ratio of an exposure measure at steady-state to that after the first dose (AI) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Half-life (T-HALF) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Effective elimination half-life that explains the degree of accumulation observed for a specific exposure measure (T-HALF eff) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab
Best overall response (BOR) | Up to two years
  To assess the preliminary anti-tumor activity
Duration of response (DOR) | Up to two years
  To assess the preliminary anti-tumor activity
Incidence of anti-drug antibody (ADA) | Up to two years
  To characterize immunogenicity
Incidence of AEs leading to discontinuation | Up to two years
  To assess the safety and tolerability of lirilumab in combination with nivolumab and ipilimumab
Maximum serum observed concentration (Cmax) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Time of maximum observed serum concentration (Tmax) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration [AUC(0-T)] | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Trough observed serum concentration (Ctrough) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Area under the serum concentration-time curve in one dosing interval [AUC(TAU)] | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Clearance (CL) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Volume of distribution at steady state (Vss) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Ratio of an exposure measure at steady-state to that after the first dose (AI) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Half-life (T-HALF) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab
Effective elimination half-life that explains the degree of accumulation observed for a specific exposure measure (T-HALF eff) | Up to two years
  To characterize the PK of lirilumab given in combination with nivolumab and ipilimumab

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Kobe, Hyōgo

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm